CLINICAL TRIAL: NCT04225104
Title: Effects of Yogic Breathing on Microvascular Endothelial Function and Symptoms in Participants With IBS
Brief Title: Yogic Breathing and IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6275
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-03

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Members of the investigative team will be blinded to the participant's group assignment until all testing is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yogic breathing intervention (Experimental): Participants assigned to this group will complete a 20-minute yogic breathing video at least 5 days per week for 4 weeks. All sessions except the initial yogic breathing session will be completed at home. Participants will complete the first session at Texas State under the supervision of the investigative team for familiarization.
  Interventions: Behavioral: Yogic breathing intervention
- Control (No Intervention): Participants in the control group will be asked to maintain their current daily activities and will be given access to the yogic breathing video once all follow-up testing has been completed at the end of week 4.

INTERVENTIONS:
Behavioral: Yogic breathing intervention — Yogic breathing will be completed while following a video provided by the investigative team. Breathing practices consist of slow, deep, relaxation breathing and are led by a certified yoga instructor.
  Arms: Yogic breathing intervention

SUMMARY:
Adults with irritable bowel syndrome (IBS) are being randomized to a yogic breathing or control condition. Participants randomized to the yogic breathing group will be asked to complete a 2-minute yogic breathing video 5 to 7 days per week at home for 4 weeks and control group participants will be asked to maintain their current activities. Participants in this group will be given access to the yogic breathing video at the end of the 4-week control period. IBS symptoms and autonomic and vascular function will be assessed at baseline and at the end of week 4 in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Must have a formal diagnosis of IBS and not be enrolled in any other clinical trials.

Exclusion Criteria:

* 1) current, regular practice of yogic breathing at least 5 minutes per day and 2) chronic obstructive pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
IBS Symptoms | Once at baseline
  IBS-Symptom Severity Scale will be administered.
IBS Symptoms | Once at the end of week 2
  IBS-Symptom Severity Scale will be administered.
IBS Symptoms | Once at the end of week 4
  IBS-Symptom Severity Scale will be administered.
Autonomic function | Once at baseline
  Heart rate variability will be assessed.
Autonomic function | Once at the end of week 2
  Heart rate variability will be assessed.
Autonomic function | Once at the end of week 4
  Heart rate variability will be assessed.
Autonomic function | Once at baseline
  Exercise heart rate recovery will be measured.
Autonomic function | Once at the end of week 2
  Exercise heart rate recovery will be measured.
Autonomic function | Once at the end of week 4
  Exercise heart rate recovery will be measured.
Microvascular function | Once at baseline
  Laser Doppler flowmetry at baseline and in response to local heating will be measured.
Microvascular function | Once at the end of week 4
  Laser Doppler flowmetry and in response to local heating will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy D Hunter, PhD, Principal Investigator — Texas State University
Locations (1):
- Stacy Hunter, San Marcos, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katherine Jurek M, Seavey H, Guidry M, Slomka E, Hunter SD. The effects of slow deep breathing on microvascular and autonomic function and symptoms in adults with irritable bowel syndrome: A pilot study. Neurogastroenterol Motil. 2022 May;34(5):e14275. doi: 10.1111/nmo.14275. Epub 2021 Oct 1. PMID 34595801